CLINICAL TRIAL: NCT01045928
Title: Phase I/II Trial of Maintenance Therapy With Lenalidomide and Rituximab Following High-Dose Chemotherapy and Autologous Stem Cell Transplantation for B-cell Non-Hodgkin Lymphoma
Brief Title: Lenalidomide And Rituximab as Maintenance Therapy in Treating Patients With B-Cell Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Extreme toxicity in Phase I, study did not proceed to Phase II
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2409; NCI-2009-01580 (Other: NCI/CTRP); CASE2409 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Adult Non-Hodgkin Lymphoma; Adult Grade III Lymphomatoid Granulomatosis; Contiguous Stage II Adult Burkitt Lymphoma; Contiguous Stage II Adult Diffuse Large Cell Lymphoma; Contiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Contiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Contiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Contiguous Stage II Adult Lymphoblastic Lymphoma; Contiguous Stage II Grade 1 Follicular Lymphoma; Contiguous Stage II Grade 2 Follicular Lymphoma; Contiguous Stage II Grade 3 Follicular Lymphoma; Contiguous Stage II Mantle Cell Lymphoma; Contiguous Stage II Marginal Zone Lymphoma; Contiguous Stage II Small Lymphocytic Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Adult Burkitt Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Noncontiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Noncontiguous Stage II Adult Lymphoblastic Lymphoma; Noncontiguous Stage II Grade 1 Follicular Lymphoma; Noncontiguous Stage II Grade 2 Follicular Lymphoma; Noncontiguous Stage II Grade 3 Follicular Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Noncontiguous Stage II Marginal Zone Lymphoma; Noncontiguous Stage II Small Lymphocytic Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Splenic Marginal Zone Lymphoma; Stage I Adult Burkitt Lymphoma; Stage I Adult Diffuse Large Cell Lymphoma; Stage I Adult Diffuse Mixed Cell Lymphoma; Stage I Adult Diffuse Small Cleaved Cell Lymphoma; Stage I Adult Immunoblastic Large Cell Lymphoma; Stage I Adult Lymphoblastic Lymphoma; Stage I Grade 1 Follicular Lymphoma; Stage I Grade 2 Follicular Lymphoma; Stage I Grade 3 Follicular Lymphoma; Stage I Mantle Cell Lymphoma; Stage I Marginal Zone Lymphoma; Stage I Small Lymphocytic Lymphoma; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Small Lymphocytic Lymphoma; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — Lenalidomide; Rituximab; Polymerase Chain Reaction; Base Sequence; Amplified Fragment Length Polymorphism Analysis; Flow Cytometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive oral lenalidomide once daily on days 1-21 and rituximab IV on day 1of courses 1, 3, 5, 7, 9, and 11.
  Interventions: Drug: lenalidomide; Biological: rituximab; Genetic: polymerase chain reaction; Genetic: nucleic acid sequencing; Genetic: polymorphism analysis; Other: flow cytometry; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: lenalidomide — Given orally
  Other Names: CC-5013; IMiD-1; Revlimid
Biological: rituximab — Given IV
  Other Names: C2B8 Monoclonal Antibody; IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Genetic: polymerase chain reaction — Correlative study
  Other Names: PCR
Genetic: nucleic acid sequencing — Correlative study
  Other Names: Gene Sequencing; Molecular Biology, Nucleic Acid Sequencing
Genetic: polymorphism analysis — Correlative study
Other: flow cytometry — Correlative study
Other: laboratory biomarker analysis — Correlative study

SUMMARY:
RATIONALE: Lenalidomide may stop the growth of cancer by blocking blood flow to the tumor. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving lenalidomide together with rituximab may be an effective treatment for B-cell non-Hodgkin lymphoma.

PURPOSE: This phase I/II trial is studying the side effects and best dose of lenalidomide when given together with rituximab as maintenance therapy in treating patients with B-cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
The study was originally intended to be Phase I/Phase II but it terminated early because of toxicity of treatment and therefore never moved to the Phase II portion of the study.

PRIMARY OBJECTIVES: I. To establish the maximum tolerated dose (MTD) and safety of lenalidomide in combination with rituximab in subjects with B-cell NHL following ASCT. (Phase I) II. To evaluate the tolerability of maintenance therapy with lenalidomide and rituximab after ASCT in subjects with B-cell NHL. (Phase II)

SECONDARY OBJECTIVES: I. To evaluate the progression-free survival of subjects with B-cell NHL receiving maintenance therapy with lenalidomide and rituximab after ASCT. II. To examine whether potential effects of lenalidomide and rituximab on progression-free survival after ASCT, compared with historical controls, vary according to histologic subtype of B-cell NHL. III. To correlate potential associations between peripheral blood levels of lymphocyte subsets including NK, T, and B cells and progression-free survival after ASCT in enrolled subjects. IV. To evaluate potential associations between progression-free survival after ASCT and polymorphisms at position 158 of FCgammaRIIIa receptor in enrolled subjects.

OUTLINE: Patients receive oral lenalidomide once daily on days 1-21of all courses and rituximab IV on day 1of courses 1, 3, 5, 7, 9, and 11. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed periodically for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form
* Able to adhere to the study visit schedule and other protocol requirements
* Histologic diagnosis of CD20+ B-cell NHL including diffuse large B-cell lymphoma, follicular lymphoma, mantle cell lymphoma and other B-cell lymphomas excluding chronic lymphocytic leukemia
* Received high-dose chemotherapy with autologous stem cell transplantation (ASCT) from 42 to 128 days before enrollment with stable disease, partial response or complete response following ASCT
* All previous cancer therapy, including radiation, hormonal therapy and surgery, must have been discontinued at least 4 weeks prior to treatment in this study
* ECOG performance status of =< 2 at study entry; Karnofsky performance status of >= 70% at study entry
* Absolute neutrophil count >= 1,500/mm^3
* Platelet count >= 75,000/mm^3
* Serum creatinine =< 2.0 mg/dL
* Phase I subjects must have estimated or measured creatinine clearance >= 60 ml/min
* Phase II subjects must have estimated or measured creatinine clearance >= 30 ml/min
* Total bilirubin =< 1.5 mg/dL
* AST (SGOT) and ALT (SGPT) =< 2 x ULN or =< 5 x ULN if hepatic metastases are present
* Disease free of prior malignancies for >= 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "insitu" of the cervix or breast
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of prescribing lenalidomide for cycle 1 (prescriptions must be filled within 7 days)
* Must also either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide
* FCBP must also agree to ongoing pregnancy testing
* Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (subjects intolerant to ASA may use warfarin or low molecular weight heparin)
* All study participants must be registered into the mandatory RevAssist program, and be willing and able to comply with the requirements of RevAssist

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that in the opinion of the investigator would prevent the subject from providing written informed consent
* Pregnant or breast feeding females (lactating females must agree not to breast feed while taking lenalidomide)
* Use of any other experimental drug or therapy within 28 days of baseline
* Known hypersensitivity to thalidomide
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
* Known hypersensitivity to rituximab
* Concurrent use of other anti-cancer agents or treatments
* Known positive for HIV or infectious hepatitis, type B or C
* Residual grade 3 or grade 4 non-hematologic toxicity after ASCT
* Transfusion requirement (red blood cells or platelets) within 14 days prior to baseline
* Use of hematopoietic growth factor (including filgrastim, pegfilgrastim, sargramostim, erythropoietin, or darbepoetin) within 14 days prior to baseline
* Any other condition not defined above, including the presence of laboratory abnormalities, which in the opinion of the investigator would place the subject at unacceptable risk if he/she were to participate in the study, or would confound the ability to interpret data from the study
* Prior use of lenalidomide either concurrently with rituximab or within 8 weeks following a dose of rituximab
* Concomitant use of other anti-cancer therapies, including radiation, thalidomide, or other investigational agents is not permitted while subjects are receiving protocol therapy during the treatment phase of the study
* Corticosteroid therapy also is not permitted while subjects are receiving protocol therapy during the treatment phase of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-01; Primary Completion 2011-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of lenalidomide (Phase I) | 24 months
Proportion of subjects who are able to complete 12 cycles of maintenance therapy with lenalidomide and rituximab after autologous stem cell transplantation (ASCT)(PHASE II) | 1 year

SECONDARY OUTCOMES:
Progression-free survival after ASCT | 24 months
Evaluation of potential differences in effects of lenalidomide and rituximab on progression-free survival after ASCT according to histologic subtypes of B-cell NHL | 24 months
Overall response rate associated with treatment with lenalidomide and rituximab after ASCT, defined as the proportion of subjects with measurable disease at enrollment who achieve a partial response or complete response | 6-12 months
Enumeration of peripheral blood lymphocyte subsets by flow cytometry, including T cells, B cells, and NK cells and analysis of potential associations between these levels with progression-free survival | At study entry, 1 month, and 1 year
Analysis of FCgammaRIIIa receptor sequences in enrolled subjects to determine the presence or absence of FCgammaRIIIa-158 polymorphisms (V/V, V/F, and F/F); determining potential associations of these polymorphisms with progression-free survival | 12 months
Incidence of non-relapse mortality (NRM) defined as death from any cause other than B-cell NHL | At 6 and 12 months
Incidence of unacceptable toxicity during study treatment | At 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dean, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Fairview Cancer Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio